CLINICAL TRIAL: NCT04358822
Title: Hemodynamic Effects of Delayed Umbilical Cord Clamping in Full-term Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dr. Reem Mahmoud, Associate Professor of Pediatrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MS-305-2019
Record Dates: First submitted 2020-04-18; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Cardiac Output, High; Cardiac Output, Low
MeSH Terms: conditions — Cardiac Output, High; Cardiac Output, Low | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30 second cord clamping (Active Comparator): Infants in this group will receive delayed cord clamping for 30 seconds.
  Interventions: Procedure: Delayed cord clamping
- 120 second cord clamping (Active Comparator): Infants in this group will receive delayed cord clamping for 120 seconds.
  Interventions: Procedure: Delayed cord clamping

INTERVENTIONS:
Procedure: Delayed cord clamping — The umbilical cord will be clamped after specific time intervals

SUMMARY:
The sequence of events at the time of delivery includes delivery of the infant, clamping of the umbilical cord, and lastly delivery of the placenta. There are some benefits for delayed cord clamping. This study aims to compare the effects of two different duration of delayed cord clamping.

Infants will be randomized into two groups based on the duration of delayed cord clamping: 30 seconds vs 120 seconds. Different hemodynamic effects will be measured in each group at different time intervals. The hypothesis of the study is that delayed cord clamping for 120 seconds is associated with better cardiac output and with other hemodynamic advantages.

DETAILED DESCRIPTION:
The study will include full term infants delivered via cesarean section. Written informed consent for participation in the study will be obtained from parents prior to delivery. Newborns will be randomly assigned into two groups according to the duration of cord clamping: Group 1: the cord will be clamped at 30 seconds, and Group 2: the cord will be clamped at 120 seconds of life. Stopwatch will be started when infants buttocks (or head if breech) are delivered from the uterus. The time elapsed will be counted aloud by the investigator in 10-second intervals. During this time, the infant will be held in linen on the mothers legs. Care will be taken not to apply traction on the cord. Milking of the cord will not be allowed. Immediately after resuscitation, infants will be attached to the leads of the electrical cardiometry device. Device output will be imported at 5, 10, and 15 minutes after birth in both groups. A follow up measurement will be imported later at 24 hours of age. In addition, a peripheral blood sample will be obtained at 24 hours of age for assessment of hemoglobin, glucose and bilirubin concentrations. .

The calculated sample size is 31 newborns in each group. This number will be adequate to detect an effect size of 10% in the mean cardiac output between the two groups with 95% confidence and 80% power. The study plans to recruit 34 infants in each group (10% attrition rate).

ELIGIBILITY:
Inclusion Criteria:

* Normal full term newborns ≥37 weeks gestational age
* Both genders are included
* Singleton
* Delivered by elective cesarean section due to previous cesarean section, cephalo-pelvic disproportion, or mal-presentation
* Successfully transitioned without need for respiratory or medication support

Exclusion Criteria:

* Neonates needing any active resuscitation
* In-utero fetal distress
* Suspected perinatal asphyxia
* Major congenital malformations
* Twin or multiple gestation
* Intrauterine growth restriction
* Placenta previa
* Mothers with cardiac disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Cardiac output | at 15 minutes
  Data imported from the electrical cardiometry device
Stroke volume | at 15 minutes
  Data imported from the electrical cardiometry device
Cardiac index | at 15 minutes
  Data imported from the electrical cardiometry device
Index of contractility | at 15 minutes
  Data imported from the electrical cardiometry device
Heart rate | at 15 minutes
  Data imported from the electrical cardiometry device
Oxygen saturation | at 15 minutes
  Data imported from the electrical cardiometry device

SECONDARY OUTCOMES:
Hemoglobin concentration | At 24 hours
  Blood sample will be obtained an analyzed
Serum glucose concentration | At 24 hours
  Blood sample will be obtained an analyzed
Serum bilirubin concentration | At 24 hours
  Blood sample will be obtained an analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Reem Mahmoud, Principal Investigator — Cairo University Children's Hospital
Locations (1):
- Cairo University Children's Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katheria AC, Wozniak M, Harari D, Arnell K, Petruzzelli D, Finer NN. Measuring cardiac changes using electrical impedance during delayed cord clamping: a feasibility trial. Matern Health Neonatol Perinatol. 2015 May 22;1:15. doi: 10.1186/s40748-015-0016-3. eCollection 2015. PMID 27057332
- [Background] Chopra A, Thakur A, Garg P, Kler N, Gujral K. Early versus delayed cord clamping in small for gestational age infants and iron stores at 3 months of age - a randomized controlled trial. BMC Pediatr. 2018 Jul 18;18(1):234. doi: 10.1186/s12887-018-1214-8. PMID 30021580
- [Background] Hsu KH, Wu TW, Wang YC, Lim WH, Lee CC, Lien R. Hemodynamic reference for neonates of different age and weight: a pilot study with electrical cardiometry. J Perinatol. 2016 Jun;36(6):481-5. doi: 10.1038/jp.2016.2. Epub 2016 Feb 18. PMID 26890553
- [Background] Mercer JS, Erickson-Owens DA, Collins J, Barcelos MO, Parker AB, Padbury JF. Effects of delayed cord clamping on residual placental blood volume, hemoglobin and bilirubin levels in term infants: a randomized controlled trial. J Perinatol. 2017 Mar;37(3):260-264. doi: 10.1038/jp.2016.222. Epub 2016 Dec 8. PMID 27929530
- [Derived] Soliman RM, Elgendy MM, Said RN, Shaarawy BI, Helal OM, Aly H. A Randomized Controlled Trial of a 30- versus a 120-Second Delay in Cord Clamping after Term Birth. Am J Perinatol. 2024 Apr;41(6):739-746. doi: 10.1055/a-1772-4543. Epub 2022 Feb 15. PMID 35170013